CLINICAL TRIAL: NCT02950129
Title: IRB-HSR # 14073 Investigation of Pelvic Girdle Dysfunction in the Low Back Pain Population
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Robin Hamill-Ruth, MD, Attending Anesthesiologist, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 14073
Record Dates: First submitted 2011-08-09; First posted 2016-10-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2011-08

CONDITIONS: Back Pain
Keywords: pelvic girdle dysfunction
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- measurements of gait (Other): all subjects will undergo 6 tests to assess gait before and after SIJ; SIJ pain diagnostic tests
  Interventions: Other: SIJ pain diagnostic tests

INTERVENTIONS:
Other: SIJ pain diagnostic tests — The subjects will undergo a specific physical exam of tests reported to be diagnostic of sacroiliac joint (SIJ) pain prior to receiving the routine injection in the SIJ; all tests will be repeated after the SIJ injection
  Other Names: back pain

SUMMARY:
The subjects will undergo a specific physical exam of tests reported to be diagnostic of sacroiliac joint (SIJ) pain prior to receiving the routine injection in the SIJ that which is being performed as part of their normal medical care. Routine care involves use of any number of these tests, but doesn't routinely include assessment of all 6 tests in all patient's treatment. The subject will fill out a Visual Analog Scale for pain and a pain drawing prior to and after the injection.

The tests will be repeated after the injection.

The investigators propose to investigate a cluster of tests proposed by Laslett as well as compare the results of the ASLR and the Gillet Test both before and after SIJ injection to determine the validity of these tests in a low back patients presenting for injections thought to be from the sacroiliac joint. The secondary purpose would be the development of a clinical predictor rule to determine examination characteristics of patients who may benefit from intraarticular injections of the SIJ.

DETAILED DESCRIPTION:
Low back pain has been the subject of extensive research in the past 10 years. Some of the efforts have focused on the effectiveness of diagnostic testing in determining the etiology of low back pain. One component of low back pain clinically can be sacroiliac joint (SIJ) dysfunction. The prevalence of sacroiliac pain in the low back pain population is reported to be approximately 10 to 30%. The diagnosis of sacroiliac pain has been an area of controversy in the literature with poor inter-tester and intra-rater reliability described for motion testing. More recently, a cluster of provocation tests has been described as predictive of the diagnosis of sacroiliac dysfunction. Laslett et al suggested that SI pain provocation tests used in examination should include a cluster of six tests. When three or more out of six tests or any two of four selected tests are positive, that showed the best predictive power in diagnosing SIJ pain. The "gold standard" for diagnosing SIJ pain in this study was pain relief with intra-articular local anesthetic block injection. When all six provocation tests do not provoke the patient's typical pain, the SIJ can be ruled out as a source of current low back pain.

Pelvic girdle pain including SIJ dysfunction has been investigated in post partum populations. The Active Straight Leg Raise (ASLR) has been shown to be reliable in post partum pelvic pain. This test is thought to help assess hypermobility in the SIJ. This test has a positive likelihood ratio (+LR)= 14.5 and a negative likelihood ratio (-LR)= .14 which indicates that this is a good test to rule in or rule out pelvic girdle pain in pregnancy. This test is thought to help assess dysfunction of the SIJ. The Gillet test has recently been reported to indicate abnormal biomechanics on the stance side by Hungerford et al. Increased hamstring activation on the stance leg has been identified as indicative of abnormal SI motion. These two tests (ASLR and Gillet) are thought to be reflective of SIJ instability or abnormal movement in, respectively, pregnancy or low back patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for sacroiliac injection with pain suspected from the sacroiliac joint

Exclusion Criteria:

* Pregnancy, allergy to contrast, inability to cooperate with screening tests, inability to understand the consent, either due to language barrier, or cognitive limitations, age > 64 years, inability to position themselves on the fluoro table for the procedure

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2009-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Predictive values of 6 tests to assess gait parameters | Day one (after SIJ injection)
  Sensitivity, specificity, positive and negative predictive values will be calculated for each SIJ pain diagnostic test using values collected prior to and following the SIJ injection

SECONDARY OUTCOMES:
Visual Analog Scale for pain | Day one (before and after SIJ injection)
  the subject will fill out a Visual Analog Scale for pain before and after the SIJ injection

CONTACTS AND LOCATIONS:
Overall Officials: Robin Hamill-Ruth, MD, Principal Investigator — UVA Anesthesiology
Locations (1):
- UVA Pain Management Center, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Broadhurst NA, Bond MJ. Pain provocation tests for the assessment of sacroiliac joint dysfunction. J Spinal Disord. 1998 Aug;11(4):341-5. PMID 9726305
- [Background] Cibulka MT, Koldehoff R. Clinical usefulness of a cluster of sacroiliac joint tests in patients with and without low back pain. J Orthop Sports Phys Ther. 1999 Feb;29(2):83-9; discussion 90-2. doi: 10.2519/jospt.1999.29.2.83. PMID 10322583
- [Background] Cibulka MT. Understanding sacroiliac joint movement as a guide to the management of a patient with unilateral low back pain. Man Ther. 2002 Nov;7(4):215-21. doi: 10.1054/math.2002.0474. No abstract available. PMID 12481788
- [Background] Hungerford B, Gilleard W, Hodges P. Evidence of altered lumbopelvic muscle recruitment in the presence of sacroiliac joint pain. Spine (Phila Pa 1976). 2003 Jul 15;28(14):1593-600. PMID 12865851
- [Background] Hungerford B, Gilleard W, Lee D. Altered patterns of pelvic bone motion determined in subjects with posterior pelvic pain using skin markers. Clin Biomech (Bristol). 2004 Jun;19(5):456-64. doi: 10.1016/j.clinbiomech.2004.02.004. PMID 15182980
- [Background] Kokmeyer DJ, Van der Wurff P, Aufdemkampe G, Fickenscher TC. The reliability of multitest regimens with sacroiliac pain provocation tests. J Manipulative Physiol Ther. 2002 Jan;25(1):42-8. doi: 10.1067/mmt.2002.120418. PMID 11898017
- [Background] Laslett M, Williams M. The reliability of selected pain provocation tests for sacroiliac joint pathology. Spine (Phila Pa 1976). 1994 Jun 1;19(11):1243-9. doi: 10.1097/00007632-199405310-00009. PMID 8073316
- [Background] Laslett M. The value of the physical examination in diagnosis of painful sacroiliac joint pathologies. Spine (Phila Pa 1976). 1998 Apr 15;23(8):962-4. doi: 10.1097/00007632-199804150-00029. No abstract available. PMID 9580969
- [Background] Laslett M, Young SB, Aprill CN, McDonald B. Diagnosing painful sacroiliac joints: A validity study of a McKenzie evaluation and sacroiliac provocation tests. Aust J Physiother. 2003;49(2):89-97. doi: 10.1016/s0004-9514(14)60125-2. PMID 12775204
- [Background] Laslett M, Aprill CN, McDonald B, Young SB. Diagnosis of sacroiliac joint pain: validity of individual provocation tests and composites of tests. Man Ther. 2005 Aug;10(3):207-18. doi: 10.1016/j.math.2005.01.003. PMID 16038856
- [Background] Laslett M, McDonald B, Tropp H, Aprill CN, Oberg B. Agreement between diagnoses reached by clinical examination and available reference standards: a prospective study of 216 patients with lumbopelvic pain. BMC Musculoskelet Disord. 2005 Jun 9;6:28. doi: 10.1186/1471-2474-6-28. PMID 15943873
- [Background] Mens JM, Vleeming A, Snijders CJ, Stam HJ, Ginai AZ. The active straight leg raising test and mobility of the pelvic joints. Eur Spine J. 1999;8(6):468-73. doi: 10.1007/s005860050206. PMID 10664304
- [Background] Mens JM, Vleeming A, Snijders CJ, Koes BW, Stam HJ. Reliability and validity of the active straight leg raise test in posterior pelvic pain since pregnancy. Spine (Phila Pa 1976). 2001 May 15;26(10):1167-71. doi: 10.1097/00007632-200105150-00015. PMID 11413432
- [Background] Mens JM, Vleeming A, Snijders CJ, Koes BW, Stam HJ. Validity of the active straight leg raise test for measuring disease severity in patients with posterior pelvic pain after pregnancy. Spine (Phila Pa 1976). 2002 Jan 15;27(2):196-200. doi: 10.1097/00007632-200201150-00015. PMID 11805667